CLINICAL TRIAL: NCT05771831
Title: Feasibility and Safety of Thrombosomes® on Time to Hemostasis in Patients Undergoing Emergency Surgery for Thoracic Aortic Dissections - a Randomized, Controlled, Open-label Investigator-initiated Pilot Trial
Brief Title: Thrombosomes® in Acute Thoracic Aortic Dissections
Acronym: TTAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jakob Stensballe, MD, PhD (Other)
Collaborators: Cellphire Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jakob Stensballe, MD, PhD, Head of research, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22061913
Record Dates: First submitted 2023-02-15; First posted 2023-03-16 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Aortic Dissection
Keywords: Surgery; Bleeding
MeSH Terms: conditions — Dissection, Thoracic Aorta; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Parallel groups, patients entering in either intervention arm or standard treatment
Masking Description: Open label treatment. Only statistician performing the data analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Thrombosomes® (Experimental): Thrombosomes® (TBX®) up to 3 doses
  Interventions: Biological: Thrombosomes®
- Standard platelet concentrate (Active Comparator): Standard platelet concentrate up to 3 doses
  Interventions: Biological: Standard platelet concentrate

INTERVENTIONS:
Biological: Thrombosomes® — The intervention with TBX® is to be administered as an intravenous infusion as hemostatic blood product as part of the Massive Transfusion Protocol (MTP).
  Other Names: TBX®; Freeze-dried platelets
  Arms: Thrombosomes®
Biological: Standard platelet concentrate — The administration of standard platelets is administrated, as part of the Massive Transfusion Protocol (MTP).
  Other Names: stPC
  Arms: Standard platelet concentrate

SUMMARY:
The hypothesis is that administration of Thrombosomes® (TBX®) as hemostatic support when terminating the cardiopulmonary bypass (CPB) in patients undergoing emergency surgery for acute thoracic aortic dissection (aTAD) is safe and least as effective when compared to standard Platelet Concentrates (stPC).

DETAILED DESCRIPTION:
The study is designed as an exploratory phase 2a, single-center randomized, controlled pilot investigator-initiated trial of administration of Thrombosomes® (TBX®) versus standard platelet concentrates (stPC) in 20 aTAD patients per arm. The patients will be enrolled in the study over a period of 15 months.

TBX® is a novel, human platelet (thrombocyte) derived lyophilized (freeze dried) hemostatic blood product for treatment of bleeding due to thrombocytopenia, dysfunctional platelet disorders or platelet consumption.

The patients will be randomized to administration of either TBX®, or stPC, as part of the Massive Transfusion Protocol (MTP) at the time of termination of the cardiopulmonary bypass (CPB) in addition to standard goal-directed hemostatic optimization based on results from thrombelastography (TEG).

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for emergency surgery on cardiopulmonary bypass pump for acute thoracic aortic dissections
* Age ≥ 18 years

Exclusion Criteria:

* Documented refusal of blood transfusion
* Aortic dissection due to trauma
* Withdrawal from active therapy
* Known hypersensitivity to TBX: the active substance, any of the excipients
* Pregnancy (non-pregnancy confirmed by patient being postmenopausal (women >55 years of age) or having a negative urine-hCG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis during surgery | During procedure
  Defined by initiation of chest closure (temporary or final closure), the placement of the first sternal wire or wound vac (ioban or film), from administration of full dose protamine.

SECONDARY OUTCOMES:
Bleeding during surgery | During procedure
  Bleeding during surgery as measured by suction, cell salvage, chest tubes, mediastinal drains, extracorporeal circulation (ECC), and in the field of surgery
Bleeding in chest tubes and mediastinal drainages on arrival in the ICU | Average 3 hours
  Volume of bleeding in chest tubes and mediastinal drains from end of surgery to arrival in the Intensive Care Unit (ICU)
Bleeding in mL in chest tube and mediastinal drainage at 24 hour after arrival in the ICU | 24 hours
  Volume of bleeding in chest tubes and mediastinal drainages from arrival in the ICU to 24 hours after ICU arrival, measured in mL
Bleeding in mL/kg in chest tube and mediastinal drainage at 24 hour after arrival in the ICU | 24 hours
  Volume of bleeding in chest tubes and mediastinal drainages from arrival in the ICU to 24 hours after ICU arrival, measured in mL/kg
Total number of blood product use during surgery | During procedure
  Number of blood products (RBC, fresh-frozen plasma (FFP), standard platelets (PLT) concentrate and/or Thrombosomes®) throughout the operation and prior to arrival at the ICU
Total volume of blood product use during surgery | During procedure
  Volume of blood products (RBC, fresh-frozen plasma (FFP), standard platelets (PLT) concentrate and/or Thrombosomes®) throughout the operation and prior to arrival at the ICU
Total number of blood product use during the first 24 hours in the ICU | 24 hours
  Numbers of blood products (RBC, FFP, standard PLT) during the first 24 hours in the ICU
Total units of blood product use during the first 24 hours in the ICU | 24 hours
  Units of blood products (RBC, FFP, standard PLT) during the first 24 hours in the ICU
Number of patients needing re-do surgery due to hemorrhage | 24 hours
  Number of patients with need for re-do surgery due to hemorrhage in the first 24 hours postoperatively
Sequential Organ Failure Assessment (SOFA) score during stay in ICU within 12 days | 12 days
  Sequential Organ Failure Assessment (SOFA) score during stay in ICU within 12 days, or until discharge from ICU, whichever comes first. Scale from 0 to 20 with 20 signifying severe organ failure
Hemostatic product use during surgery | During procedure
  Use of hemostatic products (fibrinogen concentrate, cryoprecipitate, recombinant factor VIIa) during surgery
Vasopressor free days within 30 days | 30 days
  Numbers of vasopressor free days in the ICU within 30 days
Ventilator free days | 30 days
  Numbers of ventilator free days in the ICU within 30 days
Renal replacement free days | 30 days
  Numbers of renal replacement free days in the ICU within 30 days
Length of stay in ICU | 30 days
  Numbers of days in the ICU
Length of stay in hospital | 30 days
  Numbers of days in the hospital
Mortality | 30 days
  30-day mortality after intervention
Symptomatic thrombo-embolic events | 30 days
  Numbers of symptomatic thrombo-embolic events within 30 days after intervention
Serious adverse reactions/events | 12 days
  Number of serious adverse reactions/events within the first 12 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Annette Ulrich, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No